CLINICAL TRIAL: NCT00865683
Title: DHA, Inflammation, and Insulin Sensitivity
Brief Title: DHA Supplements to Improve Insulin Sensitivity in Obese Pregnant Women (The Omega-3 Pregnancy Study)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Office of Research on Women's Health (ORWH) (NIH); Mead Johnson Nutrition (Industry); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Debra A. Krummel, PhD, RD, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 618; HL093532-01
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Overweight and Obesity; Insulin Resistance; Diabetes, Gestational; Hypertension in Pregnancy; Pre-Eclampsia
Keywords: Gestational Diabetes; Pregnancy; Docosahexaenoic Acid; DHA; Maternal-Fetal Exchange
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Diabetes, Gestational; Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Participants will receive DHA supplements.
  Interventions: Dietary Supplement: DHA Supplements
- 2 (Placebo Comparator): Participants will receive placebo capsules of corn oil.
  Interventions: Dietary Supplement: Placebo Supplements

INTERVENTIONS:
Dietary Supplement: DHA Supplements — Participants will receive 800 mg of DHA each day for approximately 3 months (until they give birth).
  Arms: 1
Dietary Supplement: Placebo Supplements — Participants will receive placebo supplements each day for approximately 3 months (until they give birth).
  Arms: 2

SUMMARY:
Women with excess adiposity while pregnant are more likely to develop gestational diabetes and high blood pressure during pregnancy than women of healthy weights. This may occur because overweight and obese pregnant women are less sensitive to insulin and have more inflammation than pregnant women of healthy weights. This study will examine the effect of a nutritional supplement, docosahexaenoic acid (DHA), on improving insulin sensitivity and lessening inflammation in overweight and obese pregnant women.

DETAILED DESCRIPTION:
The effects of overweight and obesity during pregnancy on maternal and child health can be serious and long lasting. Overweight and obese women are more likely to develop gestational diabetes or pre-eclampsia (high blood pressure and proteinuria) during pregnancy and type 2 diabetes and cardiovascular disease after pregnancy. Also, children born to these women have an increased risk of obesity, diabetes, and high blood pressure later in life. The increased risk of these diseases and conditions may occur because overweight and obese pregnant women have decreased insulin sensitivity and increased inflammation. The nutrient DHA is an omega-3 fatty acid that is important for brain function, the development of the central nervous system, and visual function in infants. DHA may also benefit both pregnant women and their babies by improving insulin sensitivity and decreasing inflammation, thereby decreasing the risk of gestational diabetes and pre-eclampsia during pregnancy. The purpose of this study is to evaluate the effect of DHA supplementation on insulin sensitivity, inflammation, and fetal growth in overweight and obese pregnant women.

This study will enroll women at 24 to 28 weeks of pregnancy. They will be followed until delivery. Participants will be randomly assigned to receive either DHA supplements or placebo on a daily basis until the end of their pregnancies. At a baseline study visit, a blood sample will be collected; height, weight, and skinfold thickness will be measured; and questionnaires to assess diet and medical history will be given. Participants will complete three diet recalls in the days after the visit, in which they will answer questions about their diet in the previous 24 hours. At a second study visit that will occur at 30 to 32 weeks of pregnancy, a blood sample will be collected. At a third study visit that will occur at 34 to 36 weeks of pregnancy, a blood sample will be collected and repeat body measurements will occur. Three diet recalls will then be completed, and participants will take part in a meal challenge, in which blood will be collected at different times after eating a study-provided breakfast. Researchers will review participants' medical records after the birth occurs.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pregnant body mass index greater than 25
* Singleton pregnancy
* Speaks English

Exclusion Criteria:

* High intake of DHA foods (i.e., more than 1 fish meal per week, use of DHA-fortified foods, or use of any supplements that contain DHA)
* Concurrent inflammatory, vascular, or metabolic disease, including diabetes, polycystic ovary disease, collagen vascular disease, inflammatory bowel disease, or infection
* Current or previous use of tobacco, street drugs, or medications known to affect inflammatory markers, including corticosteroids
* Excessive weight gain or loss before pregnancy (more than 20 pounds), including weight loss due to bariatric surgery
* Plans to leave the area during the study period
* Inability to travel to General Clinical Research Center

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | Measured at approximately Month 3

SECONDARY OUTCOMES:
Interleukin-6 (IL-6) | Measured at approximately Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Debra A. Krummel, PhD, RD, Principal Investigator — University of Cincinnati
Locations (1):
- General Clinical Research Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Lager S, Ramirez VI, Acosta O, Meireles C, Miller E, Gaccioli F, Rosario FJ, Gelfond JAL, Hakala K, Weintraub ST, Krummel DA, Powell TL. Docosahexaenoic Acid Supplementation in Pregnancy Modulates Placental Cellular Signaling and Nutrient Transport Capacity in Obese Women. J Clin Endocrinol Metab. 2017 Dec 1;102(12):4557-4567. doi: 10.1210/jc.2017-01384. PMID 29053802
- See also: Click here for the Omega-3 Pregnancy Study Web site — http://www.uc.edu/pregnancystudy